CLINICAL TRIAL: NCT00604318
Title: Is it Possible to Increase Quality of Life, Using Recombinant TSH Instead of Withdrawal of Thyroid Hormone Treatment, Before Iodine Uptake in Patients With Thyroid Cancer?
Brief Title: Quality of Life, Recombinant TSH (Thyrogen) and Thyroid Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Dathyrca 1; 2007-002713-39 (EudraCT Number); HB-2007-043 (Registry Identifier: Danish Etical commity); Data register 2007-41-120 (Registry Identifier: Danish Data Protection)
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Thyroid Cancer
Keywords: quality of life
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Thyrotropin Alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): To receive the placebo treatment in connection with the primary RI therapy and the T3 tablets and rh-TSH injections prior to second RI uptake measurement
  Interventions: Drug: rhTSH
- rh-TSH (Active Comparator): To continue with L-T3 and to receive rh-TSH stimulation with 0,9 mg Thyrogen® (Genzyme) x 2 days minus 1 and 2 prior to RI therapy, and following this to have placebo tablets and placebo injections with isotone NaCl prior to the RI uptake measurement 4-6 months later
  Interventions: Drug: rhTSH

INTERVENTIONS:
Drug: rhTSH — The patients will be randomised to either T3 (Liothyronine) pause related to the first radioiodine treatment and Thyrogen injection with continuing Liothyronine treatment related to the second treatment/uptake - or Thyrogen related to the first treatment and T3 pause related to the second treatment /uptake.
  Other Names: Thyrogen - GEnzyme

SUMMARY:
To evaluate quality of life in patients after 10 days pause of thyroid medication (Liothyronine) compared to treatment with recombinant TSH (Thyrogen) before radioiodine uptake and treatment in a double-blinded, randomised cross-over design.

DETAILED DESCRIPTION:
Patients with a thyroid follicular or papillary cancer referred to radioiodine treatment in oncological department . The patients after thyroidectomy will be treated with Liothyronine and this treatment will be paused 10 days before radioiodine. As a routine these patients will be re-evaluated with iodine uptake 4 months later.

The patients will be randomised to either T3 pause related to the first radioiodine treatment and Thyrogen injection (recombinant TSH) related to the second treatment/uptake - or Thyrogen related to the first treatment and T3 pause related to the second treatment /uptake.

All medication given in the 10 days period right before radioiodine treatment/uptake will be delivered to the patients and marked with a protocol number. In the period with T3 pause the patients will be given placebo tablets and an injection of saline (instead of Thyrogen) before treatment/uptake at the similar time as given the Thyrogen injection. A nurse otherwise not involved in the study will give the injection.

Patients will be evaluated by VAS, SF-36, and Eortc QLC30 (version 2.0) before radioiodine treatment and 3 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Follicular or papillary thyroid cancer

Exclusion Criteria:

* < 18 or > 75 years old
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
quality of life | month

CONTACTS AND LOCATIONS:
Overall Officials: Birte Nygaard, Md, PhD, Study Chair — dept of endocrinology,Herlev Hospital
Locations (1):
- Dept of Oncology, Herlev Hospital, Herlev, Herlev, Denmark